CLINICAL TRIAL: NCT04706390
Title: Comparison of the Immune Response to Natural COVID-19 Infection and Vaccination
Acronym: COVID19vac-1
Status: Recruiting | Type: Observational
Sponsor: University of Bergen (Other)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Principal Investigator, Rebecca Cox, Professor, University of Bergen
Other Study IDs: COVID-19vacc-1
Record Dates: First submitted 2021-01-11; First posted 2021-01-12 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Covid19
Keywords: Covid19; Vaccine; SARS-CoV-2 antibody
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood collection including cells.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Health care workers: 500-1000 health care workers prioritized for early vaccination
  Interventions: Biological: covid-19 vaccine
- prioritized patient populations: 2000 individuals in patient populations prioritized for vaccinations
  Interventions: Biological: covid-19 vaccine

INTERVENTIONS:
Biological: covid-19 vaccine — vaccination

SUMMARY:
The ongoing Coronavirus Disease 2019 (COVID-19) pandemic has been intensified by no population-based immunity to the severe acute respiratory disease coronavirus 2 (SARS-CoV2) and initially lack of effective treatments or vaccines available to mitigate the pandemic. Currently, two COVID-19 vaccines are available for vaccination in Europe through conditional marketing authorisation granted by the European Medicines Agency and further vaccine will be licensed. These vaccines have shown good vaccine efficacy in phase 3 vaccine trials. We will recruit subjects who will be prioritised for vaccination with the primary aim of comparing the immune responses after COVID-19 vaccination and natural SARS-CoV-2 infection. In Western Norway we have recruited cohorts of health care workers and patients infected with SARS-CoV-2 and will extend to COVID-19 vaccinees. Demographic, clinical data and repeated blood samples will be collected to evaluate the complications and kinetics, duration and breadth of the immune responses comparing natural infection to vaccination.

DETAILED DESCRIPTION:
The primary aim of this study is

* To compare immune responses after natural SARS-CoV-2 infection and COVID-19 vaccination The secondary aims are
* To compare the duration and breadth of antibody responses between natural infection and vaccination.
* To investigate the duration and breadth of B and T cellular responses between natural infection and vaccination.
* To evaluate the short and long term complications after natural infection and vaccination.
* To find out if previous infection skews the immune response after vaccination.
* To study reinfection after natural infection and vaccination.

ELIGIBILITY:
Inclusion Criteria:

* subjects prioritized by national vaccination program

Exclusion Criteria:

* Children
* unable or unwilling to provide informed consent

Ages: 20 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Comparator group: patients with natural SARS-CoV-2 infection Vaccine groups: Health care workers and high-risk population groups.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2021-01-12 (Actual); Primary Completion 2024-12-12 (Estimated); Study Completion 2030-12-12 (Estimated)

PRIMARY OUTCOMES:
immune responses | 2 months to 3 years
  spike antibody response to SARS-CoV-2

SECONDARY OUTCOMES:
Duration and breadth of B- cell responses | 2 months to 3 years
  compare serological and memory B cells after vaccination to natural infection
Duration and breadth of T cell responses | 2 months to 3 years
  compare T cell responses after vaccination to natural infection

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca J Cox, PhD, Principal Investigator — University of Bergen
Locations (1):
- University of Bergen, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Undecided
To be developed

REFERENCES:
- [Background] Cox RJ, Brokstad KA, Krammer F, Langeland N; Bergen COVID-19 Research Group. Seroconversion in household members of COVID-19 outpatients. Lancet Infect Dis. 2021 Feb;21(2):168. doi: 10.1016/S1473-3099(20)30466-7. Epub 2020 Jun 15. No abstract available. PMID 32553187
- [Background] Trieu MC, Bansal A, Madsen A, Zhou F, Saevik M, Vahokoski J, Brokstad KA, Krammer F, Tondel C, Mohn KGI, Blomberg B, Langeland N, Cox RJ; Bergen COVID-19 Research Group. SARS-CoV-2-Specific Neutralizing Antibody Responses in Norwegian Health Care Workers After the First Wave of COVID-19 Pandemic: A Prospective Cohort Study. J Infect Dis. 2021 Feb 24;223(4):589-599. doi: 10.1093/infdis/jiaa737. PMID 33247924
- [Derived] Bredholt G, Saevik M, Soyland H, Ueland T, Zhou F, Pathirana R, Madsen A, Vahokoski J, Lartey S, Halvorsen BE, Dahl TB, Trieu MC, Mohn KG, Brokstad KA, Aukrust P, Tondel C, Langeland N, Blomberg B, Cox RJ; Bergen COVID-19 Research Group. Three doses of Sars-CoV-2 mRNA vaccine in older adults result in similar antibody responses but reduced cellular cytokine responses relative to younger adults. Vaccine X. 2024 Sep 25;20:100564. doi: 10.1016/j.jvacx.2024.100564. eCollection 2024 Oct. PMID 39403561
- [Derived] Hansen L, Brokstad KA, Bansal A, Zhou F, Bredholt G, Onyango TB, Sandnes HH, Elyanow R, Madsen A, Trieu MC, Saevik M, Soyland H, Olofsson JS, Vahokoski J, Ertesvag NU, Fjelltveit EB, Shafiani S, Tondel C, Chapman H, Kaplan I, Mohn KGI, Langeland N, Cox RJ. Durable immune responses after BNT162b2 vaccination in home-dwelling old adults. Vaccine X. 2023 Apr;13:100262. doi: 10.1016/j.jvacx.2023.100262. Epub 2023 Jan 10. PMID 36643855